CLINICAL TRIAL: NCT01704911
Title: Determination of the Transradial Versus Transfemoral Coronary Angioplasty
Brief Title: Evaluate the Safety And Efficacy of the Transradial Coronary in Comparison With the Transfemoral Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CCRF Consulting Co., Ltd. (Other)
Collaborators: Peking University First Hospital (Other); Terumo Medical (Shanghai) Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Free Rate of Cardiac or Cerebrovascular Events; Transradial-transfemoral Coronary Interventions Comparison
Keywords: Transradial; Transfemoral; Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transradial Coronary Intervention (Experimental): Transradial Coronary Intervention
  Interventions: Procedure: Transradial Coronary Intervention; Device: Coronary Stent System
- Transfemoral Coronary Intervention (Experimental): Transfemoral Coronary Intervention
  Interventions: Procedure: Transfemoral Coronary Intervention; Device: Coronary Stent System

INTERVENTIONS:
Procedure: Transradial Coronary Intervention
  Arms: Transradial Coronary Intervention
Procedure: Transfemoral Coronary Intervention
  Arms: Transfemoral Coronary Intervention
Device: Coronary Stent System — Any kind of coronary stent system

SUMMARY:
The purpose of the DRAGON clinical trial is to evaluate the safety and efficacy of the transradial coronary intervention (TRI) in comparison with the transfemoral coronary intervention (TFI).

DETAILED DESCRIPTION:
Historically, performing PCI requires making an access to the peripheral arteries by an arterial puncture or cutting down. This may lead to the serious bleeding complications especially under the situation of dual antiplatelet therapy and/or potent anti-coagulation therapies. TRI is now widely accepted as the most promising alternative for TFI around the world. It is supposed to reduce the incidence of the serious bleeding complication during and after PCI, as well as the total medical cost. There have been several prospective randomized trials comparing the safety and efficacy between TRI and TFI, but none of them had enough power to show the statistically valid equivalence in the efficacy between TRI and TFI. In this study, investigators randomize approximately 1,700 patients into TRI or TFI. Investigators adopt the rate of major adverse cardiac events (MACCE) at 1 year as the primary efficacy endpoint for the study. Based on these rates at 1 year, the sample size for the non-inferiority analysis for the primary efficacy endpoint is calculated. Through this randomization trial, investigators can achieve the scientific evidence for the improved safety and equal efficacy of TRI compared to TFI. This trial has enough statistical power to draw the final conclusion in the debate between TRI and TFI.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age.
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits and treatment alternatives and he or his legally authorized representative provides signed informed consent prior to the randomization, as approved by the appropriate IEC.
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia).
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
* Allen test is required for suitable candidate.
* Patient must agree to undergo all protocol-required follow-up examinations.
* Patient must agree not to participate in any other clinical study within the duration of this trial.
* Target lesion must be able to be treated by using six-French guiding catheters.
* Target lesion can be de Novo or restenotic.
* The target lesion can be stable or unstable.

Exclusion Criteria:

* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure.
* Patient is receiving immunosuppression therapy or has known immunosuppressive or autoimmune disease (e.g. Human Immunodeficiency Virus, Lupus etc.).
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.
* Patient has other medical illness (e.g., cancer or congestive heart failure) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
* Female patients of childbearing potential who have refused a urine or blood pregnancy test (to be done within 7 days prior to index procedure), patients who are nursing at the time of index procedure and those patients who do not agree at the time of consent to use any approved form of birth control up to and including the follow-up at 1 year.
* The target lesion is considered not to be treated by using six-French guiding catheters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac or cerebrovascular events free rate | one year

SECONDARY OUTCOMES:
the major bleeding complication (BARC definition type 3 or 5)-free rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital, Japan; Yong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China